CLINICAL TRIAL: NCT05884541
Title: Promoting Math in Young Children: Leveraging Pediatric Clinics to Reach Underrepresented Children in Rural Communities
Acronym: MATH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1021594
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-05

CONDITIONS: Early Math Learning
Keywords: early math learning; preschool; rural

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors of PALS and REMA are masked to intervention status
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Children and parents receiving Early Math Texts (TipsbyText)
  Interventions: Other: TipsbyText Messages
- Control (No Intervention): Children and parents not receiving Early Math Texts (TipsbyText)

INTERVENTIONS:
Other: TipsbyText Messages — Texts sent to caregivers meant to increase parent child interaction around math and literacy, sent to participants 4x a week for 8 months
  Arms: Intervention

SUMMARY:
The goals of this clinical trial to examine how pediatricians prescribing early math enriching texts to the parents of their patients affects the early math skills of under-resourced pre-kindergarten-aged children in rural Oregon. The main question it aims to answer is: What is the impact of the text intervention on early math skills in preschool-aged children? Participants will be randomized to receive the early math text intervention or standard of care. Researchers will compare pre-and-post math performance between the intervention and control group.

DETAILED DESCRIPTION:
The goals of this clinical trial to examine how pediatricians prescribing early math enriching texts (TipsbyText) to parents of 3-4 year olds affects the math skills of under-resourced pre-kindergarten-aged children in rural Oregon. The main question it aims to answer is: What is the impact of the text intervention on early math skills in preschool-aged children using the Research-based Early Math Assessment (REMA-Brief)? Two secondary questions of the study are: What is the impact on child literacy using the Phonological Awareness Literacy Screening Tool (PALS-PreK) and parent confidence using the Development and Research in Early Math Education (DREME)? Participants will be randomized to receive intervention (the early math text intervention) or control (no texts). Researchers will compare pre-and-post math performance on the REMA-Brief (primary outcome), PALS-PreK (secondary child outcome) and DREME (secondary parent outcome) between the intervention and control group.

ELIGIBILITY:
Inclusion Criteria:

* Parents of participants must be at least 18 years of age
* Child must be 3 or 4 years old at the time of screening
* Child receives care at a participating Oregon Rural Practice-based Research Network (ORPRN) clinic
* Parent and child can communicate in English or Spanish
* Parent is able to give informed consent
* Child is eligible for Medicaid services

Exclusion Criteria:

* Parent is not able to receive text messages
* Parent is not able to read text messages
* Child is too ill to participate
* Parents who are unable to complete study activities
* Child has a sibling currently enrolled in the study
* Child has a developmental delay including neurodevelopmental disorders such as autism or syndromes associated with developmental delay (e.g. cerebral palsy, seizure disorders, attention deficit / hyperactivity disorder). Isolated expressive speech delay is not a developmental exclusion criteria.

Ages: 36 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in child early math skills measured by the Research-based Early Math Assessment (REMA-Brief) | baseline and month 9
  The Research-based Early Math Assessment (REMA-Brief) REMA-Brief assesses core mathematical abilities of children in PK and Transitional Kindergarten (TK) using an individual interview format, with explicit protocol and scoring procedures. Abilities are assessed according to theoretically and empirically based developmental progressions that underlie mathematical learning trajectories. The REMA Brief is a content-referenced test, built on psychological development that includes normative interpretations. There are twenty items; with a maximum possible raw score is 28. Average T score is 50. Standard deviation is 7.

SECONDARY OUTCOMES:
Change in child literacy measured by the Phonological Awareness Literacy Screening Tools (PALS-PreK) Score | baseline and month 9
  Screening Tool (PALS-PreK) Score [ Time Frame: Baseline and month 9 ]
  a. The PALS-PreK measures preschoolers' knowledge of literacy fundamentals: name writing, alphabet knowledge, sound awareness, print and word awareness, rhyme awareness, and nursery rhyme awareness. The English and Spanish PALS-PreK versions slightly differ in content, investigators used the "name writing, alphabet knowledge, beginning sound awareness and nursery rhyme awareness" and each section will be scored separately. Name writing (max 7 points), alphabet knowledge (part A: 26 max; part B 26 max), beginning sound awareness (10 point max), print and word awareness (10 point max). Composite score range is 0-76 with higher score indicating a better outcome.
Change in parent confidence teaching math and literacy by the Development and Research in Early Math Education (DREME) | baseline and month 9
  The DREME is a 17-item parent survey to assess parent confidence and beliefs regarding teaching and practicing math with their child.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime W Peterson, MD, MPH, Principal Investigator — Oregon Health and Science University; Lisa Chamberlain, MD, MPH, Principal Investigator — Stanford University; Susanna Loeb, PhD, Principal Investigator — Stanford University; Kendall Dunlop-Korsness, MPH, Study Director — Oregon Health and Science University; LeAnn Michaels, BS, Study Director — Oregon Health and Science University
Locations (1):
- Oregon Rural Practice Research Network, Portland, Oregon, United States